CLINICAL TRIAL: NCT02262091
Title: Strengthening Immunity of Prefrail and Frail Elderly by WGP
Brief Title: Immune Benefits of WGP in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12.22.NRC
Record Dates: First submitted 2013-10-08; First posted 2014-10-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2014-09

CONDITIONS: Elderly People
MeSH Terms: interventions — maltodextrin; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin; Biological: Influenza vaccine (incl. criterion)
- Food fibers (Experimental)
  Interventions: Dietary Supplement: Food fibers; Biological: Influenza vaccine (incl. criterion)

INTERVENTIONS:
Dietary Supplement: Food fibers
  Arms: Food fibers
Dietary Supplement: Maltodextrin
  Arms: Placebo group
Biological: Influenza vaccine (incl. criterion)

SUMMARY:
The aim of this research is to assess the immune enhancing property of food fibers in the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Male and female elderly volunteers equal or above age of 70
* Pre-frail and frail subjects (based on Fried's criteria)
* Willing to be vaccinated against influenza and having no contraindication to receive influenza vaccination
* Having obtained his/her (or his/her legal representative's) informed consent

Exclusion Criteria:

* Subject with a rapidly deteriorating health status (terminal, severe, or uncontrolled acute/chronic diseases)
* Allergy to eggs or influenza vaccine components.
* Subject who has received any vaccination in the last 3 months or has previously been vaccinated with the current seasonal influenza vaccine.
* Subject who is currently taking, or has taken in the last 4 weeks, or will take immune modulating medication during the study, including steroid, immune suppressive treatment.
* Subject who has taken antibiotics in the last 2 months prior to entering the study.
* Subject who is consuming regularly prebiotic and/or probiotic supplements, yogurts, and/or other dietary supplements.
* Personal or family history of Guillain-Barre syndrome
* BMI>35 kg/m2
* Subject who has received blood transfusion or had a blood donation during the last 4 weeks prior to the beginning of this study.
* Subject who cannot be expected to comply with the study procedures
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 4 weeks post-vaccination in antibody titers levels | Up to 1 month

SECONDARY OUTCOMES:
Measure of seroconversion | Up to 2 months
Measure of cytokines production | Up to 2 months 2014
Measure the occurence of clinical endpoints | Up to 2 months
Measure of seroprotection | Up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Leiter des Geriatrischen Zentrums Oldenburg (GZO), Oldenburg, Germany

REFERENCES:
- [Derived] Bauer JM, De Castro A, Bosco N, Romagny C, Diekmann R, Benyacoub J, Vidal K. Influenza vaccine response in community-dwelling German prefrail and frail individuals. Immun Ageing. 2017 Jul 6;14:17. doi: 10.1186/s12979-017-0098-z. eCollection 2017. PMID 28694834